CLINICAL TRIAL: NCT04079764
Title: Surveillance of Complex Renal Cysts - the SOCRATIC Pilot Study
Acronym: SOCRATICp
Status: Completed | Type: Observational
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: Canadian Urological Association (Industry); Kidney Cancer Canada (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-2871
Record Dates: First submitted 2019-07-18; First posted 2019-09-06 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Renal Cyst
Keywords: bosniak classification; Bosniak III cyst; Bosniak IV cyst; complex renal mass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- active surveillance: Patient with Bosniak III or IV lesion that decide to be followed under active surveillance
- Surgery: Patient with Bosniak III or IV lesion that decide to undergo a definitive treatment such as surgery

SUMMARY:
One third of individuals aged >60 years will be diagnosed with at least one renal cyst following abdominal imaging. These cystic lesions are categorized according to the Bosniak classification which categorizes cysts according to their degree of complexity and risk of malignancy. Growing evidence suggests that a significant proportion of Bosniak III and IV cysts are benign and that the malignant ones present low metastatic potential. Since renal surgery carries substantial morbidity (20%) and potential mortality (0.5%), active surveillance has gained attention as a potential tradeoff to surgery to overcome overtreatment. Therefore, prospective studies of long-term follow-up are needed to confirm the oncologic outcomes of this strategy for Bosniak III/IV cysts. We first designed a pilot study that will assess the feasibility of a subsequent larger multicenter observational study aiming to ascertain mid-term safety of active surveillance. The objectives of this pilot study are a) Determining patients and urologists buy-in and barriers to the proposed intervention; b) Collecting perceptions and concerns of patients and urologists; c)

DETAILED DESCRIPTION:
STUDY DESIGN - This is a two-arm multicenter prospective observational pilot study where patients with Bosniak III or IV choosing either active surveillance or surgery will be monitored closely. OBJECTIVES - PRIMARY Validate the feasibility issues (acceptability, recruitment rate, costs, protocol adherence and implementation of imaging central review) of an observational study on the treatments of complex cysts. SECONDARY a- Validate the inclusion and exclusion criteria in regard to the feasibility of the study; b- Validate the triggers for discontinuation of AS in terms of feasibility and safety for the patients. POPULATION - For the pilot study, the intended targeted population will be patients incidentally diagnosed with a Bosniak III or IV cysts and who opted to be managed by either surgery or active surveillance. METHODOLOGY - Upon written consent, patients will be explained the followup scheme which will consist of a semi-annual visits for 1 year. To mimic the upcoming larger study and to evaluate visit feasibility issues, the baseline and the follow-up visits will consist of the following items: blood results, CT-scan result, quality of life questionnaires and medical data. Baseline (prior to study entry) and follow-up abdominal imaging (CT/MRI) suspicious for progression will be reviewed centrally by an interventional radiologist at the CIUSSSE-CHUS, to confirm Bosniak classification.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18 years at the time of diagnosis
2. diagnosed with a Bosniak III or IV cyst
3. size of cystic component ≤7cm
4. solid component ≤2 cm in maximal diameter for Bosniak IV cysts
5. life expectancy >5 years (by physician's estimate)
6. diagnosis ≤6 months from accrual date
7. currently asymptomatic from the disease
8. deemed fit enough for surgery
9. willingness and ability to complete questionnaires in either French or English
10. able and willing to provide informed consent.

Exclusion Criteria:

1. history of a hereditary renal cancer syndrome
2. presence of polycystic kidney disease
3. systemic therapy for another malignancy within 12 months of recruitment date
4. uncontrolled medical illness including infections, hypertension, arrhythmias, heart failure, or myocardial infarction/unstable angina within 6 months that would predispose to immediate surgical therapy
5. metastatic disease or evidence of vascular or nodal disease
6. unwillingness to undergo monitoring and imaging studies
7. any contra-indication(s) to contrast-enhanced imaging (estimated glomerular filtration rate <30min/mL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients incidentally diagnosed with a Bosniak III or IV cysts and who opted to be managed by either surgery or active surveillance
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptability | at baseline (at enrollment, no longer than 6 months after diagnosis)
  defined by the number of patients that accept to be enrolled over the number of patients that were screened eligible
recruitment rate | at baseline (at enrollment, no longer than 6 months after diagnosis)
  defined by the number of patients that actually were enrolled per month per participating site
study costs | at the end of study (1 year after enrollment/signature of consent)
  defined by costs for research resources involved per patient per participating site
study compliance | at the end of study (1 year after enrollment/signature of consent)
  defined by the percentage of total deviations (missing data, missing visits or visits out of timeframe)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick O Richard, MD,MSc,FRSCS, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (3):
- Canada (3):
  - St Joseph's Healthcare, Hamilton, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Centre de recherche du Centre hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No
Upon completion of the study, the results will be published and disseminated by traditional knowledge transfer activities such as conference presentations (local, national and international meetings) and peer-reviewed manuscript publication.